CLINICAL TRIAL: NCT03487666
Title: OXEL: A Pilot Study of Immune Checkpoint or Capecitabine or Combination Therapy as Adjuvant Therapy for Triple Negative Breast Cancer With Residual Disease Following Neoadjuvant Chemotherapy
Brief Title: OXEL: Immune Checkpoint or Capecitabine or Combination Therapy as Adjuvant Therapy for TNBC With Residual Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1535
Record Dates: First submitted 2018-03-20; First posted 2018-04-04 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple Negative Breast Cancer; Nivolumab; Capecitabine
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Nivolumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Nivolumab 360 mg iv q3weeks for x 6 cycles
  Interventions: Drug: Nivolumab
- Arm B (Active Comparator): Capecitabine 1250mg/m2 bid D1-D14 q3 weeks x 6 cycles
  Interventions: Drug: Capecitabine
- Arm C (Experimental): Nivolumab 360mg iv q3weeks + Capecitabine 1250mg/m2 bid D1-D14 q3 weeks x 6 cycles
  Interventions: Drug: Nivolumab; Drug: Capecitabine

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a human programmed death receptor-1 (PD-1) antibody currently approved in different diseases.
  Other Names: Opdivo
  Arms: Arm A; Arm C
Drug: Capecitabine — Capecitabine was selected for Arm B given the recent results from CREATE-X trial and the increasing use by the community (feasibility). Importantly, available data from other scenarios indicates that capecitabine does not have immunosuppressive effects
  Other Names: Xeloda
  Arms: Arm B; Arm C

SUMMARY:
This pilot study will provide preliminary data regarding the role of PIS in predicting the benefit of immune checkpoint inhibition with or without chemotherapy for high risk patients with TNBC and residual disease after effective neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion criteria:

1. Biopsy proven TNBC:

   * ER- and PR- defined as ≤5% cells stain positive
   * HER2 negativity defined as:

     * IHC 0, 1+ without in situ hybridization (ISH) HER2/neu chromosome 17 ratio OR
     * IHC 2+ and ISH HER2/neu chromosome 17 ratio non-amplified with ratio less than 2.0 and if reported average HER2 copy number < 6 signals/cells
2. Residual disease of 1.0 cm at least of the primary tumor and/or node positive disease (at least ypN1)
3. Patients must have completed neoadjuvant chemotherapy; patients must NOT have received capecitabine as part of their neoadjuvant therapy regimen. Acceptable preoperative regimens include an anthracycline or a taxane, or both. Participants who received preoperative therapy as part of a clinical trial may enroll. Participants may not have received adjuvant chemotherapy after s urgery prior to randomization. . Carboplatin-containing neoadjuvant chemotherapy is also allowed). Patients who cannot complete all planned neoadjuvant treatment cycles for any reason are considered high risk and therefore are eligible for the study if they have residual disease.
4. Recovery of all toxicities from previous therapies to at least grade 1, except alopecia and ≤ grade 2 neuropathy which are allowed.
5. Must have completed definitive resection of primary tumor and have no evidence of unresected or metastatic disease at the time of study entry

   * Negative margins for both invasive and ductal carcinoma in situ (DCIS) are desirable, however patients with positive margins may enroll if the treatment team believes no further surgery is possible and patient has received radiotherapy; patients with margins positive for lobular carcinoma in situ (LCIS) are eligible
   * Either mastectomy or breast conserving surgery (including lumpectomy or partial mastectomy) is acceptable
   * Sentinel node biopsy post neoadjuvant chemotherapy (i.e. at the time of definitive surgery) is allowed; axillary dissection is encouraged in patients with lymph node involvement, but is not mandatory
6. ECOG PS 0-2
7. Patients must not be planning to receive concomitantly other biologic therapy, hormonal therapy, other chemotherapy, surgery or other anti-cancer therapy except radiation therapy while receiving treatment on this protocol.
8. At the time of registration (randomization), patients must have the following laboratory results (obtained within 28 days prior to registration):

   1. A serum TSH prior to registration to obtain a baseline value.
   2. Patients must have adequate bone marrow function as evidenced by all of the following:

      * ANC ≥ 1,500 microliter (mcL);
      * Platelets ≥ 100,000/mcL;
      * Hemoglobin ≥ 9 g/dL.
   3. Patients must have adequate hepatic function as evidenced by the following:

      * Total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN) (except Gilbert's Syndrome, who must have a total bilirubin < 3.0 mg/dL), and
      * SGOT (AST) or SGPT (ALT) and alkaline phosphatase ≤ 2.5 x IULN.
   4. Patients must have adequate renal function as evidenced by ONE of the following:

      * Serum creatinine ≤ IULN OR
      * Measured or calculated creatinine clearance ≥ 60 mL/min.
   5. Women of childbearing potential must have a negative urine or serum pregnancy test within 28 days prior to registration and within 24h prior to the start of nivolumab. In addition, women of childbearing potential must agree to have a pregnancy test every 4 weeks while on nivolumab.
9. Signed ICF
10. Age ≥18

Exclusion criteria:

1. Stage IV disease
2. Receipt of adjuvant chemotherapy
3. Diagnosis of other invasive cancer except for adequately treated cervix cancer or skin cancer, or more than 5 years since other diagnosis of invasive cancer without current evidence of disease
4. Previous exposure to capecitabine, fluorouracil or immunotherapy with anti-PD1, anti-PDL1, anti-CTLA4 or similar drugs.
5. Active autoimmune disease that has required systemic treatment in the past 2 years; replacement therapy is not considered a form of systemic therapy
6. TB, active hepatitis B, active hepatitis C or other active infection. Patients who have completed curative therapy for HCV are eligible. Patients with known HIV infection are eligible if they meet each of the following 3 criteria: CD4 counts ≥ 350 mm3; serum HIV viral load of < 25,000 IU/ml and treated on a stable antiretroviral regimen.
7. History of (non-infectious) pneumonitis that required steroids or evidence of active pneumonia
8. Uncontrolled disease
9. Chronic use of systemic steroids
10. Live vaccine within 30 days prior to registration.
11. Incapacity to provide consent or to follow clinical trial procedures
12. Pregnancy, lactation, or planning to be pregnant

Patients with microsatellite unstable tumors will not be excluded as immunotherapy as adjuvant therapy is not standard for these patients but we will prospective collect this data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candace Mainor, MD, Study Chair — MedStar Georgetown University Hospital
Locations (4):
- United States (4):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey

REFERENCES:
- [Derived] Toney NJ, Lynch MT, Lynce F, Mainor C, Isaacs C, Schlom J, Donahue RN. Serum analytes as predictors of disease recurrence and the duration of invasive disease-free survival in patients with triple negative breast cancer enrolled in the OXEL trial treated with immunotherapy, chemotherapy, or chemoimmunotherapy. J Immunother Cancer. 2025 Apr 23;13(4):e011379. doi: 10.1136/jitc-2024-011379. PMID 40274284
- See also: Related Info — https://www.nature.com/articles/s41467-024-46961-x#Sec2

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab (Arm A): Nivolumab 360 mg iv q3weeks for x 6 cycles
  Nivolumab: Nivolumab is a human programmed death receptor-1 (PD-1) antibody currently approved in different diseases.
- Capecitabine (Arm B): Capecitabine 1250mg/m2 bid D1-D14 q3 weeks x 6 cycles
  Capecitabine: Capecitabine was selected for Arm B given the recent results from CREATE-X trial and the increasing use by the community (feasibility). Importantly, available data from other scenarios indicates that capecitabine does not have immunosuppressive effects
- Nivolumab + Capecitabine (Arm C): Nivolumab 360mg iv q3weeks + Capecitabine 1250mg/m2 bid D1-D14 q3 weeks x 6 cycles
  Nivolumab: Nivolumab is a human programmed death receptor-1 (PD-1) antibody currently approved in different diseases.
  Capecitabine: Capecitabine was selected for Arm B given the recent results from CREATE-X trial and the increasing use by the community (feasibility). Importantly, available data from other scenarios indicates that capecitabine does not have immunosuppressive effects
Period: Overall Study
Arm/Group | Nivolumab (Arm A) | Capecitabine (Arm B) | Nivolumab + Capecitabine (Arm C)
Started | 15 | 15 | 15
Completed | 11 | 13 | 14
Not Completed | 4 | 2 | 1
Not completed — Disease progression | 4 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A- Nivolumab: Nivolumab 360 mg iv q3weeks for x 6 cycles
  Nivolumab: Nivolumab is a human programmed death receptor-1 (PD-1) antibody currently approved in different diseases.
- Arm B- Capecitabine: Capecitabine 1250mg/m2 bid D1-D14 q3 weeks x 6 cycles
  Capecitabine: Capecitabine was selected for Arm B given the recent results from CREATE-X trial and the increasing use by the community (feasibility). Importantly, available data from other scenarios indicates that capecitabine does not have immunosuppressive effects
- Arm C Nivolumab + Capecitabine: Nivolumab 360mg iv q3weeks + Capecitabine 1250mg/m2 bid D1-D14 q3 weeks x 6 cycles
  Nivolumab: Nivolumab is a human programmed death receptor-1 (PD-1) antibody currently approved in different diseases.
  Capecitabine: Capecitabine was selected for Arm B given the recent results from CREATE-X trial and the increasing use by the community (feasibility). Importantly, available data from other scenarios indicates that capecitabine does not have immunosuppressive effects
- Total: Total of all reporting groups
Arm/Group | Arm A- Nivolumab | Arm B- Capecitabine | Arm C Nivolumab + Capecitabine | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 13 | 41
  >=65 years | 1 | 1 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 15 | 45
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 14 | 13 | 13 | 40
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 2 | 6 | 7 | 15
  White | 11 | 6 | 8 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Peripheral Immunoscore (PIS) at Week 6
Description: PIS were developed using methods previously described (Farsaci, B. et al. Cancer Immunol. Res. 2016), based on tertile distribution of frequencies and ratios of peripheral immune cell subsets in patients prior to therapy. Immune subsets were calculated as a % of PBMC and sorted by frequency. Points were assigned to each subset in a given patient based on tertile distribution. For subsets with an expected positive effect on anti-tumor immunity zero (0) points were assigned to the low bin, one (1) point for the middle bin, and two (2) points if in the high bin. For subsets with an expected negative effect on anti-tumor immunity zero (0) points were assigned to the high bin, one (1) point for the middle bin, and two (2) points if in the low bin. The peripheral immunoscore for a given patient was the sum of points assigned to the individual PBMC subsets that were included within the immunoscore. Positive change means enhanced and negative change means reduced immune function.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: % Change in PIS
Arm/Group | Arm A- Nivolumab | Arm B- Capecitabine | Arm C Nivolumab + Capecitabine
Number analyzed (Participants) | 15 | 14 | 13
% Change in PIS | 30.63 [-37.5 to 175] | -21.9 [-55.56 to 14.286] | 32.285 [-57.143 to 300]

2. Secondary Outcome: Percent Change of Peripheral Immuno Score (PIS) at Week 12
Description: PISs were developed using methods previously described (Farsaci, B. et al. Cancer Immunol. Res. 2016), based on tertile distribution of frequencies and ratios of peripheral immune cell subsets in patients prior to therapy. Immune subsets were calculated as a % of PBMC and sorted by frequency. Points were assigned to each subset in a given patient based on tertile distribution. For subsets with an expected positive effect on anti-tumor immunity zero (0) points were assigned to the low bin, one (1) point for the middle bin, and two (2) points if in the high bin. For subsets with an expected negative effect on anti-tumor immunity zero (0) points were assigned to the high bin, one (1) point for the middle bin, and two (2) points if in the low bin. The peripheral immunoscore for a given patient was the sum of points assigned to the individual PBMC subsets that were included within the immunoscore. Positivie change mean enhanced and negative change means reduced immune function.
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: % Change in PIS
Arm/Group | Arm A- Nivolumab | Arm B- Capecitabine | Arm C Nivolumab + Capecitabine
Number analyzed (Participants) | 15 | 12 | 12
% Change in PIS | 33.3 [-37.5 to 175] | -16.2 [-55.6 to 50] | 18.83 [-62.5 to 275]

3. Secondary Outcome: Grade 3 and 4 Adverse Events
Description: The number of grade 3 and 4 adverse events as assessed clinically by an investigator, according to the National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.0 [NCI CTCAE v4.03]. Grade 4 adverse events were associated with worse outcomes.
Time Frame: From date of consent until 100 days after the last dose of study treatment, approximately up to 11 months
Measure: Number; unit: number of adverse events
Arm/Group | Arm A- Nivolumab | Arm B- Capecitabine | Arm C Nivolumab + Capecitabine
Number analyzed (Participants) | 14 | 15 | 15
number of adverse events
  Grade 3 Adverse Events | 2 | 8 | 3
  Grade 4 Adverse Events | 0 | 0 | 0

4. Secondary Outcome: Invasive Disease Free Survival (DRFS)
Description: iDFS was defined as the time from date of randomization to the date of first invasive disease recurrence, second invasive primary cancer (breast or not), or death from any cause.
Time Frame: 2 years
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A- Nivolumab | Arm B- Capecitabine | Arm C Nivolumab + Capecitabine
Number analyzed (Participants) | 15 | 15 | 15
Months | 16.75 [3.05 to 41.18] | 16.04 [0.52 to 37.05] | 21.37 [7.31 to 35.41]

5. Secondary Outcome: Circulating Tumor DNA
Description: Out of the patients with available ct-DNA samples at baseline, week 6 and week 12, the proportion of patients with detectable ct-DNA at the same timepoints.
Time Frame: 6 weeks and 12 weeks
Population: The number analyzed reflects those patients that had samples that were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A- Nivolumab | Arm B- Capecitabine | Arm C Nivolumab + Capecitabine
Number analyzed (Participants) | 13 | 12 | 13
Participants
  Baseline | 6 | 4 | 4
  Week 6: number analyzed (Participants) | 13 | 11 | 13
  Week 6 | 6 | 2 | 1
  Week 12: number analyzed (Participants) | 13 | 10 | 13
  Week 12 | 6 | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events collected from date of consent until 100 days after the last dose of study treatment, approximately up to 11 months. All cause mortality collected for up to 3 years after study drug discontinuation.
Arm/Group | Arm A- Nivolumab | Arm B- Capecitabine | Arm C Nivolumab + Capecitabine
All-Cause Mortality (participants affected / at risk) | 5/15 | 2/15 | 2/15
Serious Adverse Events (participants affected / at risk) | 3/15 | 0/15 | 3/15
Other Adverse Events (participants affected / at risk) | 14/15 | 15/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A- Nivolumab (N=15) | Arm B- Capecitabine (N=15) | Arm C Nivolumab + Capecitabine (N=15)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Breast infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Right middle lobe thoracotomy wedge resection
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A- Nivolumab (N=15) | Arm B- Capecitabine (N=15) | Arm C Nivolumab + Capecitabine (N=15)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3)
Hypothyroidism (Endocrine disorders) | 3 (4) | 0 (0) | 4 (5)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) — ear ringing
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Elevated eye pressure
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Light sensitivity
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 8 (16) | 7 (17)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) — Mouth soreness
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Abdominal Cramping
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Blood in stool
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Hungry
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (14) | 11 (18)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (8) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (6) | 3 (3)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 7 (11) | 5 (6) | 7 (12)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 0 (0) — Transaminitis
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 1 (1) — Lump at surgical incision
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — COVID infection
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Sinus infection
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Dermatitis radiation
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 3 (4)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 2 (2) | 3 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (8)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Sclerotic bone lesion
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — limited range of motion left arm
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — left arm pain
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (3)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 4 (6) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (3) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Bloody nasal discharge
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Shortness of breath
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5) | 0 (0) — Hyperpigmentation
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — skin nodule
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) — skin irritation under left breast
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Rash on chest
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03487666/Prot_SAP_000.pdf